CLINICAL TRIAL: NCT00703703
Title: A 3-way Cross-over, Randomized, Placebo-controlled, Double-blind, Multicenter Study to Assess Pharmacologic Effects of a 7-day Exposure to Darifenacin 15 mg o.d. and Tolterodine ER 4 mg o.d. on Cardiovascular Parameters in Healthy Subjects 50 Years of Age and Older
Brief Title: Pharmacologic Effects of Darifenacin and Tolterodine on Cardiovascular Parameters in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CDAR328A2414
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Heart rate, overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin
- 2 (Active Comparator): Tolterodine
  Interventions: Drug: Tolterodine
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darifenacin — Darifenacin tablets 15 mg once daily
  Other Names: Enablex
  Arms: 1
Drug: Tolterodine — Tolterodine extended release (ER) 4 mg once daily
  Other Names: Detrol LA
  Arms: 2
Drug: Placebo — Placebo tablet once daily
  Arms: 3

SUMMARY:
This study will evaluate the pharmacologic effects of exposure to darifenacin and tolterodine on cardiovascular parameters in healthy subjects 50 years of age and older

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females ≥ 50 years
* Body mass index equal to or greater than 18.5 kg/m2 and less than 35.0 kg/m2

Exclusion Criteria:

* Known or suspected allergy to tolterodine ER or darifenacin or their components
* Subjects with irregular day and night patterns such as night shift workers
* Significant medical problems know to affect heart rate (ie., hypertension, hypotension, history of heart failure, history of pulmonary disease, etc.)
* Medication with potential known to affect heart rate
* History of any malignancy within the past 5 years, with the exception of localized basal cell carcinoma of the skin
* Pregnant or nursing women
* Subjects with diseases such as urinary retention, gastric retention, uncontrolled narrow-angle glaucoma, severe renal insufficiency, etc.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Mean heart rate per 24 hours following exposure to darifenacin 15 mg o.d. and tolterodine ER 4 mg o.d., at baseline and Day 7 | 7 days

SECONDARY OUTCOMES:
Effects of darifenacin and tolterodine compared to placebo on mean heart rate per 24 hours, at baseline and Day 7 Effects of darifenacin, tolterodine and placebo on other cardiovascular parameters at baseline and Day 7 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (21):
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Tempe, Arizona
  - Investigative Site, Little Rock, Arkansas
  - Investigative Site, San Diego, California
  - Investigative Site, Washington D.C., District of Columbia
  - Investigative Site, Fort Myers, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Jupiter, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Overland Park, Kansas
  - Investigative Site, Topeka, Kansas
  - Investigative Site, Riverdale, Maryland
  - Investigative Site, Wellesley Hills, Massachusetts
  - Investigative Site, Springfield, Missouri
  - Investigative Site, Hackensack, New Jersey
  - Investigative Site, Burlington, North Carolina
  - Investigative Site, Greensboro, North Carolina
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Knoxville, Tennessee
  - Investigative Site, Morgantown, West Virginia